CLINICAL TRIAL: NCT01316757
Title: Phase II Trial of Carboplatin/Paclitaxel and Cetuximab, Followed by Carboplatin/Paclitaxel/Cetuximab and Erlotinib, With Correlative Studies in Patients With Metastatic or Recurrent Squamous Cell Carcinoma of the Head and Neck.
Brief Title: Carboplatin, Paclitaxel, Cetuximab, and Erlotinib Hydrochloride in Treating Patients With Metastatic or Recurrent Head and Neck Squamous Cell Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FER-HN-027; NCI-2011-00272 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA006927 (NIH)
Record Dates: First submitted 2011-03-08; First posted 2011-03-16 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2017-01

CONDITIONS: Metastatic Squamous Neck Cancer With Occult Primary Squamous Cell Carcinoma; Recurrent Metastatic Squamous Neck Cancer With Occult Primary; Recurrent Salivary Gland Cancer; Recurrent Squamous Cell Carcinoma of the Hypopharynx; Recurrent Squamous Cell Carcinoma of the Larynx; Recurrent Squamous Cell Carcinoma of the Lip and Oral Cavity; Recurrent Squamous Cell Carcinoma of the Nasopharynx; Recurrent Squamous Cell Carcinoma of the Oropharynx; Recurrent Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Recurrent Verrucous Carcinoma of the Larynx; Recurrent Verrucous Carcinoma of the Oral Cavity; Salivary Gland Squamous Cell Carcinoma; Stage IV Salivary Gland Cancer; Stage IV Squamous Cell Carcinoma of the Hypopharynx; Stage IV Squamous Cell Carcinoma of the Larynx; Stage IV Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IV Squamous Cell Carcinoma of the Nasopharynx; Stage IV Squamous Cell Carcinoma of the Oropharynx; Stage IV Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IV Verrucous Carcinoma of the Larynx; Stage IV Verrucous Carcinoma of the Oral Cavity; Tongue Cancer; Untreated Metastatic Squamous Neck Cancer With Occult Primary
MeSH Terms: conditions — Salivary Gland Neoplasms; Squamous Cell Carcinoma of Head and Neck; Tongue Neoplasms | interventions — Cetuximab; Paclitaxel; Taxes; Carboplatin; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Patients receive cetuximab IV over 60 minutes, paclitaxel IV over 1 hour, and carboplatin IV over 30 minutes on day 1. Beginning in course 2, patients also receive erlotinib hydrochloride PO QD on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: cetuximab; Drug: paclitaxel; Drug: carboplatin; Drug: erlotinib hydrochloride; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: cetuximab — Given IV
  Other Names: C225; C225 monoclonal antibody; IMC-C225; MOAB C225; monoclonal antibody C225
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
Drug: erlotinib hydrochloride — Given PO
  Other Names: CP-358,774; erlotinib; OSI-774
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well giving carboplatin, paclitaxel, cetuximab, and erlotinib hydrochloride together works in treating patients with metastatic or recurrent squamous cell head and neck cancer. Drugs used in chemotherapy, such as carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Erlotinib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving combination chemotherapy together with cetuximab and erlotinib hydrochloride may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the objective response rate when erlotinib is added to combination carboplatin/paclitaxel/cetuximab systemic therapy in metastatic/recurrent head and neck cancer.

SECONDARY OBJECTIVES:

I. Secondary endpoints will be toxicity, overall survival, and laboratory correlates to determine if epidermal growth factor receptor (EGFR) signaling is more effectively inhibited after the addition of erlotinib than it is after chemotherapy/cetuximab without erlotinib.

OUTLINE:

Patients receive cetuximab intravenously (IV) over 60 minutes, paclitaxel IV over 1 hour, and carboplatin IV over 30 minutes on day 1. Beginning in course 2, patients also receive erlotinib hydrochloride orally (PO) once daily (QD) on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Criteria:

* Histologically confirmed squamous cell carcinoma of the head and neck that is metastatic or recurrent
* No prior systemic therapy for metastatic/recurrent disease
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Prior chemotherapy in the induction, organ preservation or adjuvant setting is permitted if it was completed more than 4 months prior to enrollment on the current study
* Prior cetuximab is permitted if it was given for no more than 9 doses in combination with radiation therapy or chemoradiation therapy for initial treatment of locally advanced disease
* No prior erlotinib, gefitinib or lapatinib therapy is permitted; nor is prior exposure to any investigational EGFR or panErbB reversible or irreversible inhibitor or any prior panitumumab or investigational EGFR-directed monoclonal antibody permitted
* Hemoglobin > 9.0 G/dl
* Absolute neutrophil count (ANC) > 1500 cells/mcl
* Creatinine (Cr) < 1.8
* Total bilirubin =< the institution's upper limit of normal (ULN), aspartate aminotransferase (AST) and alanine transaminase (ALT) < 2 X ULN
* No chronic active viral infection
* No other malignancy within 3 years
* No chronic diarrheal condition
* Females should not be pregnant or breast feeding because chemotherapy may be harmful to the fetus or the nursing infant; also, the effects of erlotinib and cetuximab on the developing human fetus are unknown
* All females of childbearing potential must have a blood test or urine study within 2 weeks prior to randomization to rule out pregnancy
* Women of childbearing potential and sexually active males must use an accepted and effective method of contraception while on treatment and for three months after the completion of treatment
* Patients must have measurable disease based on Response Evaluation Criteria In Solid Tumors (RECIST); baseline measurements and evaluations must be obtained within < 4 weeks of randomization; all areas of disease should be recorded and mapped out in order to assess response and uniformity of response to therapy; disease in previously irradiated sites is considered measurable if there has been unequivocal disease progression or biopsy-proven residual carcinoma following radiation therapy; persistent disease without clear-cut progression after radiotherapy can be considered measurable if biopsy-proven at least 8 weeks after completion of radiation therapy
* Patients with a prior history of squamous cell or basal carcinoma of the skin or in situ cervical cancer must have been curatively treated; patients with a history of other prior malignancy must have been treated with curative intent and must have remained disease-free for 3 years post diagnosis
* No current peripheral neuropathy > grade 2 at time of randomization
* Patients must not have any co-existing condition that would preclude full compliance with the study
* Human immunodeficiency virus (HIV) positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with erlotinib
* Patients must have no history of allergic reaction to murine proteins
* Ability to understand and the willingness to sign a written informed consent
* Patients must not be receiving other investigational anti-cancer therapy
* Patients with brain metastases are not eligible
* Both men and women and members of all races and ethnic groups are eligible for this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-02-16 (Actual); Primary Completion 2015-04-07 (Actual); Study Completion 2017-10-03 (Actual)

PRIMARY OUTCOMES:
Objective response rate | Up to 3 years
  Complete plus partial response as determined by RECIST v 1.1

SECONDARY OUTCOMES:
Toxicity of study treatment | Up to 30 days post-treatment
  Assessed by National Cancer Institute (NCI) Common Toxicity Criteria (CTCAE) v.4.0. Proportions and 95% confidence intervals will be used.
Overall survival | Up to 3 years
  Will use Kaplan-Meier curves.
EGFR assay levels | Between courses 1 and 2
  Will use a Wilcoxon paired-sample test.
Response rates | Up to 3 years
  Proportions and 95% confidence intervals
Biomarkers related to EGFR | Between courses 1 and 2
  Will use Spearman correlations to assess the associations of the biomarkers with each other.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Bauman, MD, Principal Investigator — Fox Chase Cancer Center
Locations (3):
- United States (3):
  - Univesity of Rochester Medical Center, Rochester, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas

REFERENCES:
- [Derived] Bhatia A, Mehra R, Bauman J, Khan SA, Wei W, Neumeister V, Sandoval-Schaefer T, Alpaugh RK, Lango M, Rimm DL, Ridge JA, Burtness B. Phase II Trial of Chemotherapy, Cetuximab, and Erlotinib in Patients With Metastatic or Recurrent Squamous Cell Carcinoma of the Head and Neck. Head Neck. 2025 Sep;47(9):2373-2382. doi: 10.1002/hed.28152. Epub 2025 Apr 1. PMID 40166973